CLINICAL TRIAL: NCT05357547
Title: Serotonin-receptor Agonism in Reward Processing
Acronym: SARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SARP01
Record Dates: First submitted 2022-03-24; First posted 2022-05-03 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-04

CONDITIONS: Anhedonia
Keywords: 5HT1A receptor; Reward; Emotion; Memory; Buspirone
MeSH Terms: conditions — Anhedonia | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone (Experimental)
  Interventions: Drug: Buspirone 20mg
- Control (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Buspirone 20mg — Buspirone tablets in opaque capsule. Used as probe for 5HT1A agonism
  Arms: Buspirone
Drug: Placebo comparator — Lactose-sucrose tablets in opaque capsule
  Arms: Control

SUMMARY:
There is growing animal and human evidence for role of 5HT1A receptor agonism in treating depression and reward deficits. The next step is to translate this evidence directly into humans by characterising the effects of buspirone, as a 5HT1A agonist, on cognitive models of reward and emotional processing.

There is a paucity of behavioural evidence for the effect of 5HT1A receptor agonism, using buspirone as a probe, on primary reward processing (e.g. food), effort-based decision making or reward learning. Furthermore, the effects of 5HT1A agonism on non-emotive cognition, such as working memory, has yet to be investigated at a behavioural level in humans.

This study will characterise the effects of buspirone, as a probe for 5HT1A receptor agonism, on reward processing in human cognitive models. Furthermore it will examine its role in emotional processing and working memory. This will add to the evidence base of the neurocognitive effects of 5HT1A receptor agonism in humans, which is of relevance to the development of this as a target for future treatment development.

The study will be a double blinded, placebo controlled study involving healthy volunteers. Participants will receive a single dose of buspirone and then undergo a battery of psychometric testing to examine reward processing, emotional processing and a memory. Frequent monitoring of temperature and salivary cortisol shall be taken as surrogate markers of pre- and postsynaptic 5HT1A receptor activation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Male or female
* Body mass index in the range of 18 to 30
* Not currently taking any medications (except for contraception)

Exclusion Criteria:

* • Any current Axis 1 The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) psychiatric disorder
* Any previous episode of a severe mental illness,
* A first degree relative diagnosed with Bipolar Affective Disorder Type 1 or Schizophrenia
* Body Mass Index outside the range of 18 to 30 inclusive
* Any significant current medical condition likely to interfere with conduct of the study or analysis of data (epilepsy, renal disease, hepatic disease, myasthenia gravis, acute closed-angle glaucoma)
* Current use of psychoactive and / or medically significant medication as judged by a study medic, whether prescribed or bought over the counter (the contraceptive pill, the Depo-Provera injection or the progesterone implant will not result in exclusion)
* Past history of dependence to illicit substances, and any consumption of illicit substances in the three months prior to the study
* Currently pregnant or breast feeding
* Known lactase deficiency or any other problem absorbing lactose, galactose, or glucose
* Participation in a study using the same tasks in the last year
* Any physical (including visual and auditory) or language impairment that would make complying with the study protocol challenging. This includes any taste/olfactory disturbance e.g. secondary to Covid-19 infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Primary reward perception | On day of intervention (30 minutes pre-intervention and post-intervention (60 - 180 minutes))
  Visual Analogue Scale of anticipation of pleasure, intensity of taste and pleasure experienced when tasting one of four 4 tastes representing a primary reward stimulus processing.
Effort based reward task: | On day of intervention ( 90 - 180 minutes post intervention)
  offer acceptance based upon effort required (grip force on hand held dynamometer) to obtain outcome and success rate in expending correct amount of effort required for reward
Changes in reward sensitivity | On day of intervention (90 - 180 minutes post intervention)
  Sensitivity to reward as measured by the Probabilistic Instrumental Learning Task (Amount won, amount lost, total monetary amount earned , proportion of participants choosing the correct symbol in win and loss trials)

SECONDARY OUTCOMES:
Changes in recognition of emotional facial expressions | On day of intervention (90 - 180 minutes post intervention)
  Accuracy of emotion labels (e.g. disgusted face) assigned by participants to expressive faces which have appeared on a computer screen for a period of 500ms.
Changes in categorisation of emotional words | On day of intervention (90 - 180 minutes post intervention)
  Accuracy to categorise positive and negative descriptor words
Changes in recall of emotional words | On day of intervention (90 - 180 minutes post intervention)
  Number of words accurately recalled
Change in N-back task performance | On day of intervention (90 - 180 minutes post intervention)
  Accuracy on the N-back task
Change in Auditory Verbal Learning Task | On day of intervention (90 - 180 minutes post intervention)
  Accuracy on AVLT (number of items recalled across blocks)
Cortisol measurement | On day of intervention (30 minutes pre-intervention, at time of intervention, at 30 minute intervals thereafter)
  Salivary cortisol measurement at 30 minute intervals as surrogate of 5HT1A receptor activation
Temperature measurement | On day of intervention (30 minutes pre-intervention, at time of intervention, at 30 minute intervals thereafter)
  Temperature measurement at 30 minute intervals as surrogate of 5HT1A receptor activation
Temporal Experience of Pleasure scale (TEPS) | On screening day and testing day
  Measure of anticipatory and consummatory aspects of reward (state measure). 18 item questionnaire (10 items for anticipatory; 8 items for consummatory). Each item scored on 6 point Likert scale (1 = very false for me to 6 = very true for me).
  Lower score indicates greater anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Neurosciences building, Department of Psychiatry, Warneford hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be published as open access data on a secure repository (e.g. Open Science Framework https://osf/io/).
Supporting Information: Study Protocol, ICF
Time Frame: Indefinitely